CLINICAL TRIAL: NCT00261508
Title: Efficacy And Safety Of Risperidone In The Treatment Of Children With Autistic Disorder And Other Pervasive Developmental Disorders: A Canadian, Multicenter, Double-Blind, Placebo-Controlled Study
Brief Title: A Study of the Effectiveness and Safety of Risperidone Versus Placebo in the Treatment of Children With Autistic Disorder and Other Pervasive Developmental Disorders (PDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006106
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: DCild Development Disorders, Pervasive; Autistic Disorder; Developmental Disabilities; Asperger Syndrome; Rett Syndrome
Keywords: Risperidone; child development disorders; pervasive development disorders; autistic disorder; autism; developmental disabilities; antipsychotropic agents
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities; Asperger Syndrome; Rett Syndrome; Child Development Disorders, Pervasive | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the effectiveness of an oral solution of risperidone (an antipsychotic medication) versus placebo in the treatment of behavioral symptoms in children with Pervasive Developmental Disorders (PDD).

DETAILED DESCRIPTION:
The Pervasive Developmental Disorders (PDD) are a group of neuropsychiatric disorders, including autistic disorder, characterized by specific delays and deviance in social, communicative, and cognitive development with an onset typically in the first years in life. Children with PDD may show multiple, serious symptoms including hyperactivity, inattention, impulsive and aggressive behavior, repetitive movements or speech patterns, sleep disorders, screaming, and self-injurious behavior. Drug studies to date have suggested that different behavioral symptoms of PDDs respond to neuroleptics, such as risperidone. This is a randomized, double-blind, placebo-controlled study to evaluate the effectiveness of risperidone (0.02 to 0.06 mg/kg/day) compared with placebo in the treatment of behavioral symptoms in children 5 to 12 years of age with Pervasive Developmental Disorders (PDD). Patients receive study medication (risperidone or placebo) to be taken orally once a day at gradually increasing doses up to a maximum of 0.06 mg/kg, adjusted at weekly intervals to achieve optimal effectiveness while minimizing any intolerance to the drug. Treatment continues at the optimal dose through Week 8. A parent or caregiver evaluates the child's behavior and symptoms at scheduled office visits during the course of treatment. The primary measure of effectiveness is the change in the Irritability Subscale of the Aberrant Behavior Checklist (ABC) and other ABC subscales at end of treatment compared with baseline. Additional assessments of effectiveness include: the Nisonger Child Behavior Rating Form (N-CBRF); the Visual Analogue Scale (VAS), a measure of the patient's most disturbing symptom; and the Clinical Global Impression (CGI) of the overall severity of the disorder. Safety assessments include the incidence of adverse events throughout the study; measurement of vital signs (pulse, temperature, blood pressure), body weight, and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS) at specified intervals; clinical laboratory tests (hematology, biochemistry, urinalysis) before study initiation and at the end of treatment. The study hypothesis is that risperidone is more effective than placebo for the treatment of behavioral symptoms in children aged 5 to 12 years with Pervasive Developmental Disorders (PDD). Risperidone oral solution 1 mg/mL or placebo, taken orally, once daily. Days 1 - 2, dose is 0.01 mg/kg body weight. Days 3 - 7 dose is 0.02 mg/kg, increasing on Days 8 - 14 to 0.04 mg/kg (maximum), and 0.06 mg/kg (maximum) through 8 weeks. Dosage may be adjusted at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Pervasive Developmental Disorders (Autistic Disorder, Rett's Disorder, Childhood Disintegrative Disorder, Asperger's Disorder, or Pervasive Development Disorder not Otherwise Specified) by Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), Axis I criteria
* with a total score of >=30 on the Childhood Autism Rating Scale (CARS)
* receiving treatment as an out-patient
* healthy on the basis of a physical examination, electrocardiogram (ECG), and medical history at start of the study.

Exclusion Criteria:

* Diagnosis of schizophrenia or other psychotic disorders by DSM-IV criteria
* seizure during 3 months prior to study initiation or currently being treated with more than one anticonvulsant drug
* history of tardive dyskinesia (a complication of neuroleptic therapy involving involuntary movements of facial muscles)
* neuroleptic malignant syndrome (a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness)
* known hypersensitivity, intolerance, or unresponsiveness to risperidone.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 1999-08; Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Change in the Irritability Subscale of the Aberrant Behavior Checklist (ABC) and other ABC subscales at end of treatment compared with baseline

SECONDARY OUTCOMES:
Change from baseline to end of treatment in Nisonger Child Behavior Rating Form (N-CBRF), Visual Analogue Scale (VAS), and Clinical Global Impression (CGI); incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Shea S, Turgay A, Carroll A, Schulz M, Orlik H, Smith I, Dunbar F. Risperidone in the treatment of disruptive behavioral symptoms in children with autistic and other pervasive developmental disorders. Pediatrics. 2004 Nov;114(5):e634-41. doi: 10.1542/peds.2003-0264-F. Epub 2004 Oct 18. PMID 15492353